CLINICAL TRIAL: NCT02315443
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Determine the Efficacy and Safety of Intravenous NA-1 Initiated by Paramedics in the Field for Acute Cerebral Ischemia Within Three Hours of Symptom Onset
Brief Title: Field Randomization of Nerinetide (NA-1) Therapy in Early Responders
Acronym: FRONTIER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NoNO Inc. (Industry)
Collaborators: Brain Canada (Other); Djavad Mowafaghian Centre for Brain Health (Unknown); Canadian Stroke Network (Other); University of Calgary (Other); University of Toronto (Other); University of British Columbia (Other); Genome British Columbia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA-1-005; HC6-24-c 195121 (Other: Health Canada)
Record Dates: First submitted 2014-12-05; First posted 2014-12-11 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Acute Cerebral Ischemia
Keywords: Stroke; Ischemia; Prehospital; NA-1; Modified Rankin Scale; Haemorrhagic stroke; Transient ischemic attack; Nerinetide
MeSH Terms: conditions — Stroke; Ischemia; Hemorrhagic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nerinetide (NA-1) (Experimental): 2.60 mg/kg of nerinetide (up to a maximum dose of 270 mg) administered as a single 10 minute IV infusion using an ambulatory infusion pump early after stroke symptom onset.
  Interventions: Drug: Nerinetide (NA-1)
- Placebo (Placebo Comparator): Placebo administered as a single 10 minute IV infusion using an ambulatory infusion pump early after stroke symptom onset.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nerinetide (NA-1)
  Arms: Nerinetide (NA-1)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether nerinetide (NA-1) is effective in reducing global disability in patients with acute cerebral ischemia if administered early after symptom onset.

DETAILED DESCRIPTION:
Nerinetide (NA-1) is being developed as an emergency drug aimed at reducing global disability in patients with acute cerebral ischemia if administered early after symptom onset.

The primary objective is to determine the efficacy of nerinetide in reducing global disability in patients with acute stroke. The secondary objectives are to determine the efficacy of nerinetide in reducing functional dependence, reducing mortality rate, reducing worsening of stroke, improving neurological outcome and improving activities of daily living.

The leading safety objectives are to determine the effect of administering a target dose of 2.60 mg/kg (up to a maximum dose of 270 mg) IV infusion of nerinetide within three hours of symptom onset by paramedics in the field on serious adverse events and 90-day mortality.

This trial is a multicenter, randomized, double-blind, placebo-controlled, single dose study initiated prehospital in the ambulance. It is being conducted using Emergency Medical Services (EMS) in Canada. Subjects with suspected acute stroke will be identified in the field by trained paramedics using the approved stroke protocol in use by the local EMS system, and further screened for eligibility and approval by an on-call trial physician. The paramedics will administer the study drug. Upon arrival at the emergency department, subjects will receive standard-of-care.

An Independent Data Monitoring Committee will perform safety reviews of the clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Provisional diagnosis of acute stroke as identified by paramedics using the local stroke triage tool
* Respiratory rate 12-24 breaths per minute
* Oxygen saturation ≥ 90% on room air
* Systolic blood pressure < 90 or > 220 mmHg
* Weight 45-120 kg
* Last seen in usual state of health less than 3 hours before anticipated study drug initiation
* Independently ambulatory with or without devices prior to event
* LAMS score of 2-5 for at least 15 minutes and remains 2-5 at time of randomization

Exclusion Criteria:

* Lack of IV access
* Canadian Triage and Acuity Scale Level 1 and/or uncorrected airway, breathing or significant circulatory problem
* Blood sugar < 3 mmol/L (< 55 mg/dL)
* Seizure at onset of symptoms or observed by paramedic
* Glasgow coma score of <10
* Major head trauma in the last three months
* Recent stroke in the last three months
* Known or presumptive signs of pregnancy or breastfeeding
* Prisoner
* Long term care facility resident
* Known advance directive to not resuscitate
* Known participation in a clinical trial with an investigational drug or device within 30 days preceding this trial
* Pre-existing neurologic, psychiatric, or advanced systemic condition that would preclude obtaining the neurological or functional outcome evaluations

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) scale | 90 days
  The percentage of responders, using a sliding dichotomy on the mRS

SECONDARY OUTCOMES:
mRS shift analysis | 90 Days or the last rating
  Shift to reduced functional dependence analyzed across the whole distribution of scores on the mRS
Mortality rate | 90 Days
  A reduction in mortality as defined by event rate (proportion, expressed as a percentage)
Worsening of stroke rate | 90 Days
  A reduction in proportion of participants with worsening of stroke. Worsening of stroke is defined as progression, or hemorrhagic transformation, of the index stroke as documented in the study CRF that (i) is deemed life-threatening and/or (ii) results in increased disability as gauged by a ≥4 point increase from lowest NIHSS during hospitalization and/or (iii) results in death.
National Institutes of Health Stroke Scale (NIHSS) | 90 Days or the last rating
  Proportion of subjects with good neurological outcome, as defined by a score of 0-1 on the NIHSS
Barthel Index | 90 Days or the last rating
  Proportion of subjects with functional independence in activities of daily living, as defined by a score of ≥ 95 on the Barthel Index

CONTACTS AND LOCATIONS:
Overall Officials: Jim Christenson, M.D., Principal Investigator — University of British Columbia; Richard Swartz, M.D., Principal Investigator — Sunnybrook Health Sciences Centre
Locations (4):
- Canada (4):
  - Kelowna General Hospital, Kelowna, British Columbia
  - Royal Columbian Hospital, New Westminster, British Columbia
  - British Columbia Ambulance Service and British Columbia Emergency Health Services, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver Coastal Health, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Christenson J, Hill MD, Swartz RH, Adams C, Benavente O, Casaubon LK, Cheskes S, Ganesh A, Garman JD, Harris C, Harris DR, Heard K, Jenneson S, Kohli Y, Leroux M, Mayor-Nunez D, Medvedev G, Mehdiratta M, Morrison LJ, Ospel JM, Pennington S, Perez Y, Selchen D, Stebner A, Tallon J, Tkach A, Verbeek PR, Tymianski M. Efficacy and safety of intravenous nerinetide initiated by paramedics in the field for acute cerebral ischaemia within 3 h of symptom onset (FRONTIER): a phase 2, multicentre, randomised, double-blind, placebo-controlled study. Lancet. 2025 Feb 15;405(10478):571-582. doi: 10.1016/S0140-6736(25)00193-X. PMID 39955120
- [Derived] Fladt J, Ospel JM, Singh N, Saver JL, Fisher M, Goyal M. Optimizing Patient-Centered Stroke Care and Research in the Prehospital Setting. Stroke. 2023 Sep;54(9):2453-2460. doi: 10.1161/STROKEAHA.123.044169. Epub 2023 Aug 7. PMID 37548010